CLINICAL TRIAL: NCT07244913
Title: Therapeutic Effects of Instrument-assisted Versus Sound-assisted Soft Tissue Mobilization Among Patients With Chronic Non-specific Low Back Pain
Brief Title: Therapeutic Effects of Instrument-assisted Versus Sound-assisted Soft Tissue Mobilization in Chronic Non-specific Low Back Pain
Acronym: IASTM VS SASTM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Tahir Mahmood, PhD Scholar, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UOL/IREB/25/12/0015
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Non-Specific Low Back Pain; Pelvic Obliquity; Hamstring Flexibility; Physical Function; Disability; Lumbar Flexibility
Keywords: IASTM; SASTM; CPGS; Disability Index; Flexibility; Pelvic Obliquity; Physical Function; Hamstring Flexibility
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The treatment will be given to the patients after group allocation. A certified physical therapist will only provide intervention to the patients. The patients will be equally randomized in three groups. Group A = IASTM + Conventional (CON) Group B = SASTM + Conventional (CON) Group C = Conventional Therapy
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group A (Active Comparator): Group A (IASTM + Conventional therapy)
  Interventions: Device: IASTM; Other: Exercise
- Group B (Experimental): Group B (SASTM + Conventional)
  Interventions: Device: SASTM; Other: Exercise
- Group C (Other): Conventional therapy
  Interventions: Other: Exercise

INTERVENTIONS:
Device: SASTM — The therapist will apply sound instrument-assisted soft tissue mobilization (SASTM) with a convex plastic (Ceramic) tool (Beer JA, 2019).
  Arms: Group B
Device: IASTM — The IASTM technique contains a protocol for treatment that contains five components: i. Examination, ii. warm-up exercises 5 min iii. IASTM treatment (e.g., 30-60 seconds per session), iv. Post treatment stretching and strengthening, v. Icing (only when sub-acute inflammation is of concern).
  Arms: Group A
Other: Exercise — In conventional therapy, patients will be given an exercise program that will be targeted to low back muscles. This will be include three type of exercise focusing on stretching, strengthening and postural correction exercise.(Yana et al., 2024)

SUMMARY:
Chronic low back pain (CLBP) is the most common medical problem observed among musculoskeletal pain and spinal pain problems. It can reduce the movements due to muscular imbalances, decreased activity of daily living, and effects on health-related quality of life. It is the major cause of activity limitation, work absence, and reported clinical issues. Most of the cases of low back pain remained undiagnosed and received only symptomatic management.

DETAILED DESCRIPTION:
There is limited literature on advanced soft tissue release techniques provided by primary healthcare practitioners specific to low back pain. Some of the studies are based on soft tissue mobilization using a mechanically assisted method, but they have limited outcomes, acute effects, and small sample sizes, which limit their generalization. Further literature is limited in the comparison of IASTM and SASTM. Further, there are limited techniques that can facilitate practitioners to identify the restrictions.

Firstly, instrument-assisted soft tissue mobilization (IASTM), due to its body contour and shape, recognizes specific tissue lesions and restriction sites while targeting specific points rather than using manual methods that cover a larger contact area. Using the mechanotransduction phenomenon, its mechanical stimuli initiate biochemical signals that trigger cellular responses and ultimately functional improvement. Biomechanically, fascial elasticity, fascial stiffness, and viscosity absorb and distribute forces. While tissue hydration level is increased, that is compromised in chronic low back pain.

Secondly, sound-assisted soft tissue mobilization could be an intervention for treating musculoskeletal disorders. The SASTM technique has the potential to be a game-changer in pain management after IASTM. The sound decreases as adhesions are broken. While breakdown of scar tissue can be a facilitator for ease of movement patterns.

ELIGIBILITY:
Inclusion Criteria:

* Pain between the inferior gluteal folds and the costal margins.
* Pain with a duration of a minimum of 24 weeks.
* Moderate to severe pain (>3) was measured using the Numeric Pain Rating Scale.
* Straight Leg raise Limited (hamstring tightness)

Exclusion Criteria:

* Pain in lower back with radiating/referring but limited to proximal legs
* Pain for the last 03 months and at least half of the days in the last six months.
* Presence of neurological problem/deficit/disease (e.g., nerve root compression, motor deficit, paresthesia) and lower limb symptoms.
* Presence of disease like Infection, tumors, spondylolisthesis grade II or higher, vertebral fractures, identifiable cause like endometriosis
* Medicine like immunosuppression or steroid medication;
* Spinal deformities
* History of severe rheumatic, orthopedic, or cardiovascular disease in the last three months before study participation.
* Previously diagnosed Osteoporosis
* SIJ dysfunction is evaluated by a positive compression test.
* BMI over 35.
* Skin allergy or hypersensitivity that can lead to skin irritation due to IASTM/SASTM tools.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity will be noted at baseline ,after the 2nd week, 3rd week, 4th week, and follow up will be taken at 2nd month, and after the 4th month post intervention.
  The pain will be assessed using Chronic Pain grading Scale (CPGS).
Flexibility | The lumbar flexibility will be noted at basline after the 2nd week, 3rd week, 4th week, and follow up will be taken at 2nd month, and after the 4th month post intervention.
  Modified-Modified Schober Test will be used to measure Lumbar flexibility.

SECONDARY OUTCOMES:
Function | The functional movement screening will be noted at baseline, after the 2nd week, 3rd week, 4th week, and follow up will be taken at 2nd month, and after the 4th month post intervention.
  Functional movement Screen (FMS) will be used.
Disability | Disability will be assessed before treatment, after the 2nd month, and 4th month post-intervention.
  Roland Morris Disability Index will be used to measure disability Index.
Hamstring Flexibility | Hamstring flexibility will be measured at basline, 2nd month, and after the 4th month post intervention.
  Active knee Extension Test will be used to assess hamstring Flexibility.

OTHER OUTCOMES:
Pelvic obliquity | The pelvic obliquity will be assessed before treatment, after 2nd month and 4th month post-intervention.
  Leg length difference will be measured as an indicator of pelvic obliquity.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Arif Memorial Teaching Hospital, Lahore, Punjab Province
  - Re Active Physio Clinic Lahore., Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708
- [Background] Yilmaz Yelvar GD, Cirak Y, Dalkilinc M, Parlak Demir Y, Guner Z, Boydak A. Is physiotherapy integrated virtual walking effective on pain, function, and kinesiophobia in patients with non-specific low-back pain? Randomised controlled trial. Eur Spine J. 2017 Feb;26(2):538-545. doi: 10.1007/s00586-016-4892-7. Epub 2016 Dec 15. PMID 27981455
- [Background] Markman JD, Czerniecka-Foxx K, Khalsa PS, Hayek SM, Asher AL, Loeser JD, Chou R. AAPT Diagnostic Criteria for Chronic Low Back Pain. J Pain. 2020 Nov-Dec;21(11-12):1138-1148. doi: 10.1016/j.jpain.2020.01.008. Epub 2020 Feb 6. PMID 32036046
- [Background] Ahmed UA, Maharaj SS, Van Oosterwijck J. Effects of dynamic stabilization exercises and muscle energy technique on selected biopsychosocial outcomes for patients with chronic non-specific low back pain: a double-blind randomized controlled trial. Scand J Pain. 2021 Feb 24;21(3):495-511. doi: 10.1515/sjpain-2020-0133. Print 2021 Jul 27. PMID 33641272
- [Background] Bodes Pardo G, Lluch Girbes E, Roussel NA, Gallego Izquierdo T, Jimenez Penick V, Pecos Martin D. Pain Neurophysiology Education and Therapeutic Exercise for Patients With Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):338-347. doi: 10.1016/j.apmr.2017.10.016. Epub 2017 Nov 11. PMID 29138049
- [Background] Yana M, Gunes M, Simsek A, Apaydin AS, Akinci C, Ozmen T. The Effect of Graston Technique on Pain, Proprioception, Flexibility, and Disability in Patients with Chronic Non-specific Low Back Pain. Altern Ther Health Med. 2024 Apr;30(4):24-30. PMID 38702163
- [Background] Cheatham SW, Kreiswirth E, Baker R. Does a light pressure instrument assisted soft tissue mobilization technique modulate tactile discrimination and perceived pain in healthy individuals with DOMS? J Can Chiropr Assoc. 2019 Apr;63(1):18-25. PMID 31057174
- [Background] Brandl A, Egner C, Schwarze M, Reer R, Schmidt T, Schleip R. Immediate Effects of Instrument-Assisted Soft Tissue Mobilization on Hydration Content in Lumbar Myofascial Tissues: A Quasi-Experiment. J Clin Med. 2023 Jan 28;12(3):1009. doi: 10.3390/jcm12031009. PMID 36769657
- [Background] Brandl A, Egner C, Reer R, Schmidt T, Schleip R. Associations between Deformation of the Thoracolumbar Fascia and Activation of the Erector Spinae and Multifidus Muscle in Patients with Acute Low Back Pain and Healthy Controls: A Matched Pair Case-Control Study. Life (Basel). 2022 Oct 28;12(11):1735. doi: 10.3390/life12111735. PMID 36362889
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- See also: Sound-Assisted Soft Tissue Mobilization will be used. — https://sastm.com/pages/why-choose-sastm